CLINICAL TRIAL: NCT00493818
Title: An Open-label Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the AKT Inhibitor GSK690693 Given on Various Schedules in Subjects With Solid Tumors or Lymphoma
Brief Title: Open-label Study to Investigate the Safety, Tolerability, PK, and Pharmacodynamics of the AKT Inhibitor GSK690693
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKT106757
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Cancer
Keywords: GSK690693,; Solid Tumors,; Lymphoma,; AKT
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — GSK690693

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK690693

SUMMARY:
This study is a first time in human, Phase I, open-label study to determine recommended doses and schedules, based on maximum tolerated doses and biologically active doses, for the AKT inhibitor GSK690693.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of solid tumor malignancy or lymphoma that is not responsive to standard therapies or for which there is no approved therapy
* Female patients of child-bearing potential must be willing to abstain from intercourse from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication or be willing to consistently and correctly use an acceptable method of birth control.

Exclusion Criteria:

* Prior anti-cancer therapy within the prior 28 days.
* History of diabetes.
* Coronary artery disease/myocardial infarction, acute coronary syndromes within the past 6 months.
* Use of theophylline and warfarin within 14 days prior to the first dose of study drug.
* Current use of oral corticosteroids (note: Inhaled corticosteroids are permitted.)
* Participation in an investigational study within the prior 28 days.
* Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of GSK690693 given weekly or twice weekly over 1 - 4 hours. | given weekly or twice weekly over 1 - 4 hours

SECONDARY OUTCOMES:
Blood pressure and heart rate every 8 hours. | every 8 hours.
12-lead ECGs will be conducted at 4, 8, 10, 12, 14, 24hrs | 4, 8, 10, 12, 14, 24hrs
Pharmacokinetics and Pharmacodynamics via blood draws before, during, and after the infusion. | draws before, during, and after the infusion
Urinalysis samples while the patient is hospitalized | while the patient is hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: AKT106757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AKT106757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AKT106757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AKT106757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AKT106757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AKT106757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AKT106757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register